CLINICAL TRIAL: NCT01837537
Title: Evaluation of Respiration Rate Parameters in a Hospital Population Using a Nellcor Bedside Respiratory Patient Monitoring System With Respiration Rate Version 2.0
Brief Title: Respiration Rate V2.0 in a Hospital Setting
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0399
Record Dates: First submitted 2013-04-17; First posted 2013-04-23 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-06

CONDITIONS: Respiratory Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment: no treatment, prospective observational

SUMMARY:
The purpose of this study is to meet the respiration rate accuracy specifications for the study pulse oximeter monitoring system (study device) in a hospitalized volunteer population when compared to established technologies for measuring parameters related to respiration, such as Capnograph Respiration Rate (RR)(CO2).

DETAILED DESCRIPTION:
Volunteer subjects from a hospital setting (see specific inclusion/exclusion criteria) over the age of 18, male and female, who provide written informed consent prior to the procedure, and are without any contact skin allergies to adhesives found in standard pulse oximetry sensors. A cross section of demographics - cardiovascular, respiratory, and metabolic type cases should be considered for a broad distribution of medical and surgical patients.

The study consists of measuring parameters related to respiration in hospitalized volunteers by means of the Bedside Respiratory Patient Monitoring System with RR V2.0 (Nightingale). The production-equivalent Nightingale device and multiparameter reference devices will be attached to the subject via sensors, nasal cannulas and ECG leads and the information from all devices will be captured continuously for up to 40 minutes to allow for at least 30 minutes of artifact free data 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* 18 years or older.
* A patient at the study site on a General Care Floor or General Surgery Care Floor.
* Subject is willing and able to provide written consent.

Exclusion Criteria:

* Subject is younger than 18.
* Subject has severe contact allergies that may cause a reaction to standard adhesive materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors.
* Subject has an abnormality that may prevent proper application of the device.
* Subject is in atrial fibrillation.
* Subject has a documented history of frequent premature ventricular contractions (PVCs), defined as greater than 3 in 30 seconds or greater than 6 in 60 seconds.
* Subject has an implanted pacemaker.
* Subject is unwilling or unable to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteer subjects from a hospital setting on the general care floor or general surgical care floor
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Lumbley, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | no Treatment
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | no Treatment
Number analyzed (Participants) | 90
Age, Continuous [Mean (Full Range); unit: years] | 54.2 [18 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 76
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Mean Error (ME) +/- 1 Breath Per Minute, RR Sensor
Description: The software calculates respiration rate values via Adult Respiratory Sensor with a mean error of +/- 1 breath per minute relative to a capnography based reference. The Mean Error value estimates the mean difference in simultaneous estimates of respiration rate (the Respiration Rate calculated from the sensor and the Respiration Rate calculated from capnography).
Time Frame: up to 40 minutes of continuous monitoring
Population: 90 subjects were enrolled. Out of the 90 enrolled 75 yielded valid data. The remaining 15 subjects did not meet the predetermined data criteria (such as reference was too noisy, timing of observations could not be matched, etc.)
Measure: Mean (Standard Deviation); unit: BrPM (breaths per minute)
Arm/Group | no Treatment
Number analyzed (Participants) | 75
BrPM (breaths per minute) | -0.82 (2.19)

2. Secondary Outcome: Mean Error (ME) +/- 1 Breath Per Minute, Max-N Sensor
Description: The software calculates respiration rate values via the Max-N Sensor with a mean error of +/- 1 breath per minute relative to a capnography based reference. The Mean Error value estimates the mean difference in simultaneous estimates of respiration rate (the Respiration Rate calculated from the sensor and the Respiration Rate calculated from capnography). The error value estimates the mean difference in simultaneous estimates of respiration rate (the Respiration Rate calculated from the Max-N sensor minus the Respiration Rate calculated from capnography.
Time Frame: up to 40 minutes of continuous monitoring
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BrPM
Arm/Group | no Treatment
Number analyzed (Participants) | 75
BrPM | -0.16 (2.85)

ADVERSE EVENTS:
Arm/Group | no Treatment
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No